CLINICAL TRIAL: NCT07338084
Title: OpioidRedoxStudyII
Acronym: ORRS
Status: Not yet recruiting | Type: Observational
Sponsor: Europainclinics z.ú. (Other)
Collaborators: Pavol Jozef Safarik University (Other); F.D.Roosevelt Banska Bystrica Slovak Republic (Unknown)
Responsible Party: Sponsor
Other Study IDs: B1112025
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Oxidative Stress; Opioid Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood-derived samples, including serum and plasma, collected for the assessment of redox-related biomarkers. Samples will be retained for biochemical analyses and will not be used for DNA extraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Tramadol Cohort
- Group 2: Tapentadol Cohort
- Group 3: Buprenorphine - Morphin Cohort
- Group 4: Fentanyl Cohort

SUMMARY:
This observational study aims to examine the relationship between opioid use and redox balance in adults. Redox balance reflects the level of oxidative stress in the body, which is known to play an important role in many biological processes and diseases.

Participants who use opioids will be included in the study. No experimental treatment or changes to current medical care will be provided as part of this study. Biological samples may be collected to assess redox-related biomarkers, and relevant clinical and demographic information will be recorded.

The results of this study are expected to improve understanding of how opioid exposure is associated with redox balance in adults. This information may help inform future research on the biological effects of opioids and potential strategies to reduce harm associated with long-term opioid use.

DETAILED DESCRIPTION:
Opioids are widely used for the management of acute and chronic pain; however, prolonged opioid exposure has been associated with a range of systemic effects beyond analgesia. Increasing evidence suggests that oxidative stress and alterations in redox balance may play a role in the biological effects of opioids, potentially contributing to tissue damage, inflammation, and other adverse outcomes.

The OpioidRedoxStudy II is an observational study designed to further investigate the association between opioid use and redox balance in adults. This study builds on previous findings by focusing on redox-related biomarkers that reflect oxidative and antioxidative processes in the human body. The study does not involve any experimental intervention, randomization, or modification of participants' current medical treatment.

Participants using opioids will be assessed using biological samples collected according to the study protocol. These samples will be analyzed for markers related to redox balance. In addition, relevant clinical, demographic, and opioid exposure data will be collected to allow for exploratory analyses of associations between opioid use patterns and redox-related measures.

The primary objective of this study is to characterize the relationship between opioid exposure and redox balance in adults. Secondary objectives include exploring potential associations between redox-related biomarkers and clinical characteristics. The findings of this study are intended to contribute to a better understanding of the biological effects of opioid use and to support future research aimed at reducing opioid-related harm.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Receiving opioid therapy (tramadol, tapentadol, morphine, fentanyl, or buprenorphine) as part of routine clinical care
* Stable opioid treatment for at least a predefined minimum period prior to enrollment (according to the study protocol)
* Ability to provide written informed consent
* Ability to comply with study procedures, including blood sampling and completion of questionnaires

Exclusion Criteria:

* Acute opioid intoxication or withdrawal at the time of enrollment
* Use of investigational drugs or participation in another interventional clinical trial that could interfere with study outcomes
* Severe acute illness or unstable medical condition that, in the investigator's judgment, would interfere with study participation
* Known pregnancy or breastfeeding
* Inability to provide informed consent
* Any condition that, in the opinion of the investigator, would make participation unsafe or compromise the quality of the collected data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of adult patients receiving opioid therapy as part of routine clinical care. Participants are treated with tramadol, tapentadol, morphine, fentanyl, or buprenorphine and are enrolled into predefined observational cohorts based on the type of opioid used. The study population includes individuals with ongoing opioid exposure who are able to provide informed consent and comply with study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Redox Balance Assessed by Circulating Redox-Related Biomarkers | At baseline (at enrollment)
  Assessment of redox balance using circulating redox-related biomarkers measured in blood-derived samples. Biomarker levels will be compared across opioid exposure cohorts to evaluate associations between opioid type and redox balance.
Association Between Genetic Variants Related to Opioid Metabolism and Opioid-Related Adverse Effects | From enrollment to 12 months after enrollment
  Assessment of the association between selected genetic variants related to opioid metabolism and signaling and the occurrence of opioid-related adverse effects and treatment intolerance across opioid exposure cohorts.

SECONDARY OUTCOMES:
Chronification Risk Assessment | At baseline (at enrollment)
  Assessment of the risk of pain chronification using a validated pain chronification risk assessment questionnaire in adults receiving opioid therapy.
Pain Severity and Interference Assessed by the Brief Pain Inventory | At baseline and during follow-up up to 12 months after enrollment
  Assessment of pain severity and pain-related interference with daily activities using the Brief Pain Inventory (BPI) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pavol JoSef Safarik, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of the collected data, including genetic information and detailed clinical variables. Data sharing is further restricted to ensure participant confidentiality and compliance with applicable data protection regulations.

REFERENCES:
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Kotagal V, Pontone GM, Bohnen NI. Chronic pain and cognitive decline: exploring the link in aging and neurodegenerative disorders. Pain Med. 2015;16(3):430-442. PMCID: PMC4377400.
- [Background] Martuliak I, Golubnitschaja O, Chvala L, Kapalla M, Ferencik M, Bubeliny M, Venglarcik M, Kocan L. Pain chronification risk assessment: advanced phenotyping and scoring for prediction and treatments tailored to individualized patient profile. EPMA J. 2024 Nov 15;15(4):739-750. doi: 10.1007/s13167-024-00383-3. eCollection 2024 Dec. PMID 39635026
- [Background] Richie M, Koob GF, Schulteis G. Genetic variability in ABCB1 and analgesic response: implications for morphine efficacy. J Pain. 2018;19(10):1090-1098. doi:10.1016/j.jpain.2018.04.004.
- [Background] in W, Zhang Y, Chen D, et al. ABCB1 C3435T polymorphism affects opioid dose requirements through P-glycoprotein-mediated transport. Biomed Pharmacother. 2024;172:114007. doi:10.1016/j.biopha.2024.114007.
- [Background] Rakvag TT, Klepstad P, Baar C, Kvam TM, Dale O, Kaasa S, Krokan HE, Skorpen F. The Val158Met polymorphism of the human catechol-O-methyltransferase (COMT) gene may influence morphine requirements in cancer pain patients. Pain. 2005 Jul;116(1-2):73-8. doi: 10.1016/j.pain.2005.03.032. PMID 15927391
- [Background] Ho KYY, Loh S, Lim JF, et al. Influence of OPRM1 and COMT polymorphisms on pain perception and opioid responses: a randomized controlled trial. Pharmacogenomics J. 2020;20(6):762-769. PMCID: PMC7651441.
- [Background] Chidambaran V, Zhang X, Martin LJ, et al. Genetic predictors of postoperative respiratory depression after pediatric tonsillectomy: OPRM1 and ABCB1 variants. Pharmacogenomics J. 2015;15(5):430-435. PMID: 25349169.
- [Background] Stamer UM, Stuber F, Muders T, Musshoff F. Respiratory depression with tramadol in a patient with renal impairment and CYP2D6 gene duplication. Anesth Analg. 2008 Sep;107(3):926-9. doi: 10.1213/ane.0b013e31817b796e. PMID 18713907
- [Background] Zeng L, Zhen J, Wang T, et al. Thioredoxin-1 regulates morphine-induced addictive behavior through redox modulation in the nucleus accumbens. Front Pharmacol. 2020;11:573434. doi:10.3389/fphar.2020.573434.
- [Background] Ahmadi A, Shadboorestan A, Ahmatkesh A. Opioid administration and oxidative stress: a review of the literature. J Opioid Manag. 2017;13(1):35-44. PMID: 28296619.